CLINICAL TRIAL: NCT02040766
Title: A Randomized, Double-Blind, Double-Dummy, Placebo-Controlled, Parallel-Group, 12-Week Clinical Study to Assess the Efficacy and Safety of 80 or 160 mcg/Day of Beclomethasone Dipropionate Delivered Via Breath-Actuated Inhaler (BAI) or Metered-Dose Inhaler (MDI) in Pediatric Patients 4 Through 11 Years of Age With Persistent Asthma
Brief Title: A Safety and Efficacy Study of Beclomethasone Dipropionate Delivered Via Breath-Actuated Inhaler (BAI) or Metered-Dose Inhaler (MDI) in Participants Ages 4-11 Years Old With Persistent Asthma
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BDB-AS-302; 2013-004632-30 (EudraCT Number)
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Results first posted 2018-02-12 (Actual); Last update posted 2021-11-09 (Actual); Status verified 2021-11

CONDITIONS: Asthma
Keywords: asthma; breath-actuated inhaler; metered dose inhaler
MeSH Terms: conditions — Asthma | interventions — Beclomethasone; Albuterol; Bronchodilator Agents; Metered Dose Inhalers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- BDP 80 mcg BAI (Experimental): Beclomethasone dipropionate (BDP) was administered via a breath-actuated inhaler (BAI) twice daily (40 mcg twice a day).
  Placebo MDI twice daily for blinding.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) at 90 mcg ex-actuator) or equivalent was used as rescue medication throughout the study.
  Interventions: Drug: Beclomethasone dipropionate BAI; Drug: albuterol/salbutamol 90 mcg; Drug: Placebo MDI
- BDP 160 mcg BAI (Experimental): Beclomethasone dipropionate (BDP) was administered via a breath-actuated inhaler (BAI) twice daily (80 mcg twice a day).
  Placebo MDI twice daily for blinding.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) at 90 mcg ex-actuator) or equivalent was used as rescue medication throughout the study.
  Interventions: Drug: Beclomethasone dipropionate BAI; Drug: albuterol/salbutamol 90 mcg; Drug: Placebo MDI
- BDP 80 mcg MDI (Active Comparator): Beclomethasone dipropionate (BDP) was administered via a metered-dose inhaler (MDI) twice daily (40 mcg twice a day).
  Placebo BAI twice daily for blinding.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) at 90 mcg ex-actuator) or equivalent was used as rescue medication throughout the study.
  Interventions: Drug: Placebo BAI; Drug: albuterol/salbutamol 90 mcg; Drug: Beclomethasone dipropionate MDI
- BDP 160 mcg MDI (Active Comparator): Beclomethasone dipropionate (BDP) was administered via a metered-dose inhaler (MDI) twice daily (80 mcg twice a day).
  Placebo BAI twice daily for blinding.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) at 90 mcg ex-actuator) or equivalent was used as rescue medication throughout the study.
  Interventions: Drug: Placebo BAI; Drug: albuterol/salbutamol 90 mcg; Drug: Beclomethasone dipropionate MDI
- Placebo BAI and MDI (Placebo Comparator): Placebo was administered via breath-actuated inhaler (BAI) twice daily. Additionally placebo was administered via metered-dose inhaler (MDI) twice daily.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) at 90 mcg ex-actuator) or equivalent was used as rescue medication throughout the study.
  Interventions: Drug: Placebo BAI; Drug: albuterol/salbutamol 90 mcg; Drug: Placebo MDI

INTERVENTIONS:
Drug: Beclomethasone dipropionate BAI — Beclomethasone dipropionate (BDP), was delivered by a single inhalation using a breath-actuated inhaler (BAI) at levels of 40 mcg or 80 mcg per inhalation, twice each day.
  Other Names: BDP; breath-actuated inhaler
  Arms: BDP 160 mcg BAI; BDP 80 mcg BAI
Drug: Placebo BAI — Placebo was delivered by a single inhalation using a breath-actuated inhaler (BAI) twice each day.
  Other Names: breath-actuated inhaler
  Arms: BDP 160 mcg MDI; BDP 80 mcg MDI; Placebo BAI and MDI
Drug: albuterol/salbutamol 90 mcg — Rescue medication (albuterol/salbutamol hydrofluoroalkane (HFA) MDI [90 mcg ex-actuator] or equivalent) for use on an as-needed basis for the immediate relief of asthma symptoms throughout the treatment period.
  Other Names: bronchodilators
Drug: Beclomethasone dipropionate MDI — Beclomethasone dipropionate (BDP), was delivered by a single inhalation using a metered-dose inhaler (MDI) at levels of 40 mcg or 80 mcg per inhalation, twice each day.
  Other Names: BDP; metered-dose inhaler; QVAR®
  Arms: BDP 160 mcg MDI; BDP 80 mcg MDI
Drug: Placebo MDI — Placebo was delivered by a single inhalation using a metered-dose inhaler (MDI) twice each day.
  Arms: BDP 160 mcg BAI; BDP 80 mcg BAI; Placebo BAI and MDI

SUMMARY:
This randomized, double-blind, double-dummy, placebo-controlled, parallel-group, 12-week study will evaluate the efficacy and safety of beclomethasone dipropionate (80 or 160 mcg/day) administered via breath-actuated inhaler (BAI) and metered-dose inhaler (MDI) in pediatric patients 4 through 11 years of age with persistent asthma, compared with placebo.

Patients took 1 inhalation (with assistance from parents/guardians/caregivers, as needed) from each of 2 devices (BAI device followed by MDI device in that order) twice daily as per the double-dummy study design: 1 BAI treatment or placebo device and 1 MDI treatment or placebo device for a total of 2 inhalations each time.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Asthma diagnosis: The patient has a diagnosis of asthma as defined by the National Institute of Health (NIH). The asthma diagnosis has been present for a minimum of 3 months and has been stable (defined as no exacerbations and no changes in medication) for at least 30 days before screening visit
* Severity of disease: The patient has persistent asthma, with a forced expiratory volume in 1 second (FEV1) 40% to 90% of the value predicted for age, height, and sex at screening visit (SV)
* Current asthma therapy: The patient is currently being treated with 1 of the following: 1) a stable daily dosage of an inhaled corticosteroid (ICS) in the range of 88-176 mcg/day of fluticasone propionate (or equivalent) for a minimum of 4 weeks (28 days) before screening visit 2) a stable daily dosage of non-corticosteroid therapy 3) a daily dose of ICS plus a long-acting beta2-agonist (LABA) (at a dose less than or equivalent to fluticasone propionate 100 mcg/salmeterol 50 mcg twice daily)
* Reversibility of disease: The patient has demonstrated at least 12% reversibility of FEV1 within 30 minutes after 2-4 inhalations of albuterol/salbutamol hydrofluoroalkane (HFA) MDI (90 mcg ex-actuator) or equivalent at screening visit or on retesting.
* Other criteria apply, please contact the investigator for more information

Exclusion Criteria:

* The patient has a history of life-threatening asthma, defined for this protocol as an asthma episode that required intubation and/or was associated with hypercapnia, respiratory arrest, or hypoxic seizures.
* The patient is pregnant or lactating, or plans to become pregnant during the study period or for 30 days after the patient's last study-related visit (for eligible patients only, if applicable). Any patient becoming pregnant during the study will be withdrawn from the study.
* The patient has a known hypersensitivity to any corticosteroid or any of the excipients in the study drug or rescue medication formulation.
* The patient has used tobacco products within the past year (eg, cigarettes, cigars, chewing tobacco, or pipe tobacco, as applicable).
* The patient has had an asthma exacerbation requiring oral corticosteroids within 30 days before screening visit, or has had any hospitalization for asthma within 2 months before screening visit.
* The patient has historical or current evidence of a clinically significant disease. Significant disease is defined as any disease that in the medical judgment of the investigator would put the safety of the patient at risk through participation or that could affect the efficacy or safety analysis if the disease/condition worsened during the study.
* Other criteria apply, please contact the investigator for more information

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 628 (Actual)
Dates: Start 2013-12; Primary Completion 2016-02 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teva Medical Expert, MD, Study Director — Teva Branded Pharmaceutical Products R&D, Inc.
Locations (102):
- United States (75):
  - Teva Investigational Site 12346, Hoover, Alabama
  - Teva Investigational Site 12294, Montgomery, Alabama
  - Teva Investigational Site 10925, Phoenix, Arizona
  - Teva Investigational Site 12349, Little Rock, Arkansas
  - Teva Investigational Site 10903, Costa Mesa, California
  - Teva Investigational Site 10911, Downey, California
  - Teva Investigational Site 10901, Huntington Beach, California
  - Teva Investigational Site 12297, Huntington Beach, California
  - Teva Investigational Site 10880, Mission Viejo, California
  - Teva Investigational Site 10895, Orange, California
  - Teva Investigational Site 10924, Paramount, California
  - Teva Investigational Site 10910, Rolling Hills Estates, California
  - Teva Investigational Site 12343, Roseville, California
  - Teva Investigational Site 12298, San Diego, California
  - Teva Investigational Site 12300, San Diego, California
  - Teva Investigational Site 12295, San Jose, California
  - Teva Investigational Site 12312, West Covina, California
  - Teva Investigational Site 10937, Centennial, Colorado
  - Teva Investigational Site 10899, Colorado Springs, Colorado
  - Teva Investigational Site 10894, Aventura, Florida
  - Teva Investigational Site 12335, Gainesville, Florida
  - Teva Investigational Site 12336, Homestead, Florida
  - Teva Investigational Site 12345, Homestead, Florida
  - Teva Investigational Site 12315, Miami, Florida
  - Teva Investigational Site 12341, Miami, Florida
  - Teva Investigational Site 12342, Miami, Florida
  - Teva Investigational Site 10919, Orlando, Florida
  - Teva Investigational Site 12281, Sarasota, Florida
  - Teva Investigational Site 12332, Winter Park, Florida
  - Teva Investigational Site 10935, Gainesville, Georgia
  - Teva Investigational Site 10912, Lawrenceville, Georgia
  - Teva Investigational Site 10927, Savannah, Georgia
  - Teva Investigational Site 10885, Owensboro, Kentucky
  - Teva Investigational Site 12317, Covington, Louisiana
  - Teva Investigational Site 12296, Baltimore, Maryland
  - Teva Investigational Site 12323, White Marsh, Maryland
  - Teva Investigational Site 10897, North Dartmouth, Massachusetts
  - Teva Investigational Site 10932, Ypsilanti, Michigan
  - Teva Investigational Site 10914, Plymouth, Minnesota
  - Teva Investigational Site 10917, Columbia, Missouri
  - Teva Investigational Site 10916, Rolla, Missouri
  - Teva Investigational Site 12331, Missoula, Montana
  - Teva Investigational Site 10922, Brick, New Jersey
  - Teva Investigational Site 10909, Ocean City, New Jersey
  - Teva Investigational Site 12289, Verona, New Jersey
  - Teva Investigational Site 10939, Asheville, North Carolina
  - Teva Investigational Site 12348, Charlotte, North Carolina
  - Teva Investigational Site 10893, Raleigh, North Carolina
  - Teva Investigational Site 10888, Canton, Ohio
  - Teva Investigational Site 12302, Fairfield, Ohio
  - Teva Investigational Site 10921, Toledo, Ohio
  - Teva Investigational Site 12285, Toledo, Ohio
  - Teva Investigational Site 10906, Oklahoma City, Oklahoma
  - Teva Investigational Site 10915, Oklahoma City, Oklahoma
  - Teva Investigational Site 12314, Oklahoma City, Oklahoma
  - Teva Investigational Site 10891, Tulsa, Oklahoma
  - Teva Investigational Site 10892, Medford, Oregon
  - Teva Investigational Site 10898, Portland, Oregon
  - Teva Investigational Site 12273, Pittsburgh, Pennsylvania
  - Teva Investigational Site 12282, Warwick, Rhode Island
  - Teva Investigational Site 10902, North Charleston, South Carolina
  - Teva Investigational Site 10938, Orangeburg, South Carolina
  - Teva Investigational Site 12347, Beaumont, Texas
  - Teva Investigational Site 10926, Boerne, Texas
  - Teva Investigational Site 10908, Dallas, Texas
  - Teva Investigational Site 10918, Dallas, Texas
  - Teva Investigational Site 12291, El Paso, Texas
  - Teva Investigational Site 12329, Live Oak, Texas
  - Teva Investigational Site 10890, New Braunfels, Texas
  - Teva Investigational Site 10904, San Antonio, Texas
  - Teva Investigational Site 10929, San Antonio, Texas
  - Teva Investigational Site 10879, Waco, Texas
  - Teva Investigational Site 10883, Richmond, Virginia
  - Teva Investigational Site 10886, Bellingham, Washington
  - Teva Investigational Site 10913, Greenfield, Wisconsin
- Croatia (3):
  - Teva Investigational Site 60017, Čakovec
  - Teva Investigational Site 60018, Zagreb
  - Teva Investigational Site 60019, Zagreb
- Mexico (8):
  - Teva Investigational Site 21037, Guadalajara
  - Teva Investigational Site 21042, Guadalajara
  - Teva Investigational Site 21039, Mexico City
  - Teva Investigational Site 21045, Mexico City
  - Teva Investigational Site 21035, Monterrey
  - Teva Investigational Site 21043, San Lucas Tepetlacalco
  - Teva Investigational Site 21047, San Lucas Tepetlacalco
  - Teva Investigational Site 21051, Zapopan
- Poland (9):
  - Teva Investigational Site 53276, Bialystok
  - Teva Investigational Site 53267, Krakow
  - Teva Investigational Site 53269, Lodz
  - Teva Investigational Site 53272, Lodz
  - Teva Investigational Site 53271, Lublin
  - Teva Investigational Site 53274, Lublin
  - Teva Investigational Site 53273, Tarnów
  - Teva Investigational Site 53275, Wroclaw
  - Teva Investigational Site 53270, Zawadzkie
- Ukraine (7):
  - Teva Investigational Site 58165, Dnipropetrovsk
  - Teva Investigational Site 58171, Kharkiv
  - Teva Investigational Site 58168, Kryvyi Rih
  - Teva Investigational Site 58167, Kyiv
  - Teva Investigational Site 58172, Kyiv
  - Teva Investigational Site 58169, Zaporizhzhia
  - Teva Investigational Site 58170, Zaporizhzhya

REFERENCES:
- [Result] Vandewalker M, Hickey L, Small CJ. Efficacy and safety of beclomethasone dipropionate breath-actuated or metered-dose inhaler in pediatric patients with asthma. Allergy Asthma Proc. 2017 Sep 14;38(5):354-364. doi: 10.2500/aap.2017.38.4078. Epub 2017 Jul 14. PMID 28710850

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were screened at 123 centers in Croatia, Mexico, Poland, Ukraine, and the United States. The intent-to-treat (ITT) population included all randomly assigned patients
Pre-assignment Details: Patients were randomly assigned to treatment through a qualified randomization service provider. This system was used to ensure a balance across treatment groups, within each stratum
Period: Overall Study
Arm/Group | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI
Started | 127 | 126 | 125 | 125 | 125
Completed | 109 | 116 | 113 | 112 | 112
Not Completed | 18 | 10 | 12 | 13 | 13
Not completed — Adverse Event | 1 | 1 | 1 | 0 | 2
Not completed — Withdrawal by Subject | 4 | 3 | 2 | 3 | 2
Not completed — Non-compliance | 0 | 1 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 1 | 2 | 3 | 0
Not completed — Lost to Follow-up | 4 | 1 | 3 | 1 | 4
Not completed — Not reported | 1 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 6 | 3 | 4 | 6 | 5

BASELINE CHARACTERISTICS:
Population: Intent to treat (ITT) population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI | Total
Number analyzed (Participants) | 127 | 126 | 125 | 125 | 125 | 628
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (2.06) | 8.5 (2.10) | 8.4 (1.24) | 8.2 (1.78) | 8.4 (1.86) | 8.3 (1.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 52 | 46 | 49 | 50 | 238
  Male | 86 | 74 | 79 | 76 | 75 | 390
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 4 | 4 | 3 | 1 | 15
  Asian | 0 | 2 | 2 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 42 | 34 | 33 | 37 | 49 | 195
  White | 71 | 69 | 69 | 76 | 63 | 348
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 11 | 17 | 17 | 9 | 12 | 66

OUTCOME MEASURES:

1. Primary Outcome: Standardized Baseline-adjusted Trough Morning Percent Predicted Forced Expiratory Volume in 1 Second (FEV1) Area Under the Effect Curve From Time 0 to 12 Weeks (AUEC(0-12wk))
Description: Trough morning FEV1 measurements were taken pre-dose and pre-rescue bronchodilator treatment for asthma. Baseline was defined as baseline trough morning percent predicted FEV1. Pulmonary function measurements (including FEV1) were obtained electronically by spirometry. All pulmonary function test data were submitted to a central reading center for evaluation. The highest ('best attempt') FEV1 value from 3 acceptable and 2 repeatable maneuvers (maximum of 8 attempts) was used.
Time Frame: Day 1 (baseline), Weeks 2, 4, 8, 12
Population: The full analysis set (FAS) included all patients in the ITT population who received at least 1 dose of study drug and had at least 1 post baseline trough morning (pre-dose and pre-rescue bronchodilator) assessment of percent predicted FEV1.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI
Number analyzed (Participants) | 113 | 111 | 116 | 114 | 114
liters | 2.62 (0.744) | 5.43 (0.742) | 3.25 (0.732) | 3.54 (0.734) | 3.71 (0.734)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 80 mcg BAI; ANCOVA model with effects due to baseline trough morning percent predicted FEV1, sex, age, current protocol-allowed asthma therapy (inhaled corticosteroid (ICS) or non-corticosteroid (NCS) therapy) at the time of screening visit, during the run-in period, and during treatment; Test type: Superiority; p = 0.0063, ANCOVA — significance at 0.05; Mean Difference (Final Values) = 2.81, 95% CI 2-sided [0.796 to 4.821]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 160 mcg BAI; ANCOVA model with effects due to baseline trough morning percent predicted FEV1, sex, age, current protocol-allowed asthma therapy (ICS or NCS therapy) at the time of screening visit, during the run-in period, and during treatment; Test type: Superiority; p = 0.5332, ANCOVA — significance at 0.05; Mean Difference (Final Values) = 0.63, 95% CI 2-sided [-1.354 to 2.614]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 80 mcg MDI; [analysis description as in outcome 1, analysis 2]; Test type: Superiority; p = 0.3649, ANCOVA — significance at 0.05; Mean Difference (Final Values) = 0.92, 95% CI 2-sided [-1.077 to 2.924]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 160 mcg MDI; Test type: Superiority; p = 0.2823, ANCOVA; Mean Difference (Final Values) = 1.09, 95% CI 2-sided [-0.902 to 3.088]

2. Secondary Outcome: Change From Baseline in Weekly Average of Daily Trough Morning Peak Expiratory Flow (PEF) Over the 12-week Treatment Period
Description: The analysis of change from baseline in weekly average of daily trough morning (pre-dose and pre-rescue bronchodilator) PEF calculated across the 12-week treatment period was performed using a mixed model for repeated measures (MMRM) with effects due to baseline weekly average of daily trough morning PEF.
Time Frame: Day 1 (baseline), weeks 1-12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI
Number analyzed (Participants) | 124 | 124 | 122 | 121 | 123
liters | 4.3 (2.11) | 15.6 (2.08) | 12.8 (2.12) | 11.9 (2.11) | 10.8 (2.11)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 80 mcg BAI; Test type: Superiority; p = 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 11.3, 95% CI 2-sided [5.58 to 17.06]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 160 mcg BAI; Test type: Superiority; p = 0.0041, Mixed Models Analysis; Mean Difference (Final Values) = 8.5, 95% CI 2-sided [2.71 to 14.24]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 80 mcg MDI; Test type: Superiority; p = 0.0103, Mixed Models Analysis; Mean Difference (Final Values) = 7.6, 95% CI 2-sided [1.79 to 13.35]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 160 mcg MDI; Test type: Superiority; p = 0.0278, Mixed Models Analysis; Mean Difference (Final Values) = 6.5, 95% CI 2-sided [0.71 to 12.23]

3. Secondary Outcome: Change From Baseline in Weekly Average of Daily Evening Peak Expiratory Flow (PEF) Over the 12-week Treatment Period
Description: The analysis of change from baseline in the weekly average of daily evening PEF across the 12-week treatment period was performed using a mixed model for repeated measures (MMRM) with effects due to baseline weekly average of daily evening PEF.
Time Frame: Day 1 (baseline), weeks 1-12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI
Number analyzed (Participants) | 124 | 124 | 122 | 121 | 123
liters | 1.4 (2.11) | 13.1 (2.09) | 11.4 (2.12) | 11.3 (2.12) | 10.1 (2.12)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 80 mcg BAI; Test type: Superiority; p < 0.0001, Mixed Models Analysis; Mean Difference (Final Values) = 11.7, 95% CI 2-sided [5.96 to 17.45]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 160 mcg BAI; Test type: Superiority; p = 0.0007, Mixed Models Analysis; Mean Difference (Final Values) = 10.0, 95% CI 2-sided [4.20 to 15.76]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 80 mcg MDI; Test type: Superiority; p = 0.0008, Mixed Models Analysis; Mean Difference (Final Values) = 9.9, 95% CI 2-sided [4.11 to 15.68]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 160 mcg MDI; Test type: Superiority; p = 0.0031, Mixed Models Analysis; Mean Difference (Final Values) = 8.7, 95% CI 2-sided [2.95 to 14.49]

4. Secondary Outcome: Change From Baseline in the Weekly Average of Total Daily (24-hour) Use of Albuterol/Salbutamol Inhalation Aerosol (Number of Inhalations) Over Weeks 1-12
Description: The change from baseline in the weekly average of total daily (24-hour) use of albuterol/ salbutamol inhalation aerosol (number of inhalations) across the 12 weeks was analyzed using a mixed model for repeated measures (MMRM).
Time Frame: Day 1 (baseline), weeks 1-12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: Number of inhalations
Arm/Group | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI
Number analyzed (Participants) | 124 | 124 | 122 | 121 | 123
Number of inhalations | -0.36 (0.069) | -0.72 (0.068) | -0.50 (0.069) | -0.41 (0.069) | -0.54 (0.069)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 80 mcg BAI; Test type: Superiority; p = 0.0002, Mixed Models Analysis; Mean Difference (Final Values) = -0.36, 95% CI 2-sided [-0.548 to -0.174]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 160 mcg BAI; Test type: Superiority; p = 0.1320, Mixed Models Analysis; Mean Difference (Final Values) = -0.14, 95% CI 2-sided [-0.331 to 0.044]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 80 mcg MDI; Test type: Superiority; p = 0.5866, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.240 to 0.136]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 160 mcg MDI; Test type: Superiority; p = 0.0587, Mixed Models Analysis; Mean Difference (Final Values) = -0.18, 95% CI 2-sided [-0.369 to 0.007]

5. Secondary Outcome: Change From Baseline in the Weekly Average of the Total Daily Asthma Symptom Score Over Weeks 1-12
Description: The total daily asthma symptom score is the average of the daytime and nighttime scores analyzed using an mixed model for repeated measures (MMRM). Baseline was defined as the average of recorded morning and evening asthma symptom scores over the 7 days before randomization. Daytime Scores range from 0=No symptoms during the day to 5=Symptoms so severe that I could not go to work or perform normal daily activities; Nighttime Scores range from 0=No symptoms during the night to 4=Symptoms so severe that I did not sleep at all. The daily asthma symptom score was therefore 0 - 9 with 0=no symptoms during the day or night and 9=severe symptoms both day and night.
Time Frame: Day 1 (baseline), weeks 1-12
Population: Full analysis set
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI
Number analyzed (Participants) | 124 | 124 | 122 | 121 | 123
units on a scale | -0.27 (0.036) | -0.44 (0.036) | -0.36 (0.036) | -0.31 (0.036) | -0.36 (0.036)
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 80 mcg BAI; Test type: Superiority; p = 0.0011, Mixed Models Analysis; Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.261 to -0.065]
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 160 mcg BAI; Test type: Superiority; p = 0.0869, Mixed Models Analysis; Mean Difference (Final Values) = -0.09, 95% CI 2-sided [-0.185 to 0.013]
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 80 mcg MDI; Test type: Superiority; p = 0.4388, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.138 to 0.060]
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 160 mcg MDI; Test type: Superiority; p = 0.1041, Mixed Models Analysis; Mean Difference (Final Values) = -0.08, 95% CI 2-sided [-0.180 to 0.017]

6. Secondary Outcome: Kaplan-Meier Estimates For Time to Withdrawal Due to Meeting Stopping Criteria for Worsening Asthma During the 12-week Treatment Period
Description: Time to withdrawal due to meeting stopping criteria was defined as number of days elapsed from the date of first dose of double-blind study treatment to the date of withdrawal due to meeting stopping criteria.
  Kaplan-Meier estimates (median and 95% CI of the median) are not applicable if the proportion of participants withdrawn is less than 0.5.
Time Frame: Day 1 to 12 weeks
Population: Full analysis set
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI
Number analyzed (Participants) | 124 | 124 | 122 | 121 | 123
Days | NA [NA to NA] — Too few participants withdrew to calculate estimate. | NA [NA to NA] — Too few participants withdrew to calculate estimate. | NA [NA to NA] — Too few participants withdrew to calculate estimate. | NA [NA to NA] — Too few participants withdrew to calculate estimate. | NA [NA to NA] — Too few participants withdrew to calculate estimate.
Statistical Analysis 1: Comparison: Placebo BAI and MDI vs BDP 80 mcg BAI; Test type: Superiority; p = 0.2870, Log Rank
Statistical Analysis 2: Comparison: Placebo BAI and MDI vs BDP 160 mcg BAI; Test type: Superiority; p = 0.5257, Log Rank
Statistical Analysis 3: Comparison: Placebo BAI and MDI vs BDP 80 mcg MDI; Test type: Superiority; p = 0.9982, Log Rank
Statistical Analysis 4: Comparison: Placebo BAI and MDI vs BDP 160 mcg MDI; Test type: Superiority; p = 0.7633, Log Rank

ADVERSE EVENTS:
Time Frame: - Run-In: Days -21 to Day 0 - Double-blind Study Treatment: Day 1 to Week 12
Description: Run-In Placebo arm includes participants who were randomized.
Groups:
- Run-in Placebo: Placebo was administered via breath-actuated inhaler (BAI) twice daily. Additionally placebo was administered via metered-dose inhaler (MDI) twice daily. Both were single-blind therapies giving participants experience with the devices.
  Prestudy asthma medications were adjusted according to the protocol.
  Albuterol/salbutamol hydrofluoroalkane (HFA) metered-dose inhaler (MDI) at 90 mcg ex-actuator) or equivalent was used as rescue medication throughout the study.
Arm/Group | Run-in Placebo | Placebo BAI and MDI | BDP 80 mcg BAI | BDP 160 mcg BAI | BDP 80 mcg MDI | BDP 160 mcg MDI
Serious Adverse Events (participants affected / at risk) | 0/628 | 0/127 | 0/126 | 0/125 | 0/125 | 0/125
Other Adverse Events (participants affected / at risk) | 1/628 | 8/127 | 6/126 | 13/125 | 15/125 | 11/125
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Run-in Placebo (N=628) | Placebo BAI and MDI (N=127) | BDP 80 mcg BAI (N=126) | BDP 160 mcg BAI (N=125) | BDP 80 mcg MDI (N=125) | BDP 160 mcg MDI (N=125)
Nasopharyngitis (Infections and infestations) | 0 (0) | 4 (5) | 5 (6) | 11 (14) | 6 (7) | 6 (7)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (7) | 1 (1) | 3 (3) | 9 (11) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has the right 60 days before submission for publication to review/provide comments. If the Sponsor's review shows that potentially patentable subject matter would be disclosed, publication or public disclosure shall be delayed for up to 90 additional days in order for the Sponsor, or Sponsor's designees, to file the necessary patent applications. In multicenter trials, each PI will postpone single center publications until after disclosure or publication of multicenter data.